CLINICAL TRIAL: NCT03444922
Title: Effects of Oral Ingestion of BPA on Insulin and Glucose Responses
Brief Title: Effects of BPA on Insulin and Glucose Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Todd Hagobian, Associate Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPJune62018
Record Dates: First submitted 2018-02-08; First posted 2018-02-26 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Environmental Exposure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Double-blinded study; Study statistician computer generated randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants consume Vanilla Wafer cookie
  Interventions: Other: Placebo
- BPA 4 ug/kg BW (Experimental): Participants consume 4 ug/kg BW of BPA on a Vanilla Wafer Cookie
  Interventions: Other: BPA 4 ug/kg BW
- BPA 50 ug/kg BW (Experimental): Participants consume 50 ug/kg BW of BPA on a Vanilla Wafer Cookie
  Interventions: Other: BPA 50 ug/kg BW

INTERVENTIONS:
Other: Placebo — Ingestion of Placebo
  Arms: Placebo
Other: BPA 4 ug/kg BW — Oral BPA ingestion of 4 ug/kg BW
  Arms: BPA 4 ug/kg BW
Other: BPA 50 ug/kg BW — Oral BPA ingestion of 50 ug/kg BW
  Arms: BPA 50 ug/kg BW

SUMMARY:
The National Institutes of Health has encouraged research examining effects of BPA, yet evidence in humans evaluating the effects of BPA on insulin and glucose concentrations remains exclusively associative in nature. Thus, the primary purpose of this study is to determine whether an acute oral ingestion of BPA impacts insulin and glucose concentrations, and other endocrine factors (Pro-insulin, C-Peptide, Estrogen, triglycerides). Findings from this pilot study will inform public health recommendations for food packaging and provide much needed experimental evidence as to whether BPA poses any public health risk.

DETAILED DESCRIPTION:
The prevalence of diabetes is well established affecting >29 million Americans with 90-95% of these individuals diagnosed with type 2 diabetes. The etiology of type 2 diabetes is not fully understood, but clearly diet, physical activity, and genetics play roles. Emerging data suggests a novel hypothesis that synthetic non-persistent endocrine disruptors used in a variety of common consumer goods, including the industry-produced chemical bisphenol A (BPA) play a pivotal role in type 2 diabetes and obesity rates. In support of this hypothesis, National Health and Nutrition Examination Survey (NHANES), Nurses' Health Study II (NHSII), and other cross-sectional data have shown associations between urinary BPA concentrations and type-2 diabetes, pre-diabetes, insulin resistance, and hemoglobin A1c. The National Institutes of Health has encouraged research examining effects of BPA, yet evidence in humans evaluating the effects of BPA on insulin and glucose concentrations remains exclusively associative in nature. Thus, the primary purpose of this study is to determine whether an acute oral ingestion of BPA impacts insulin and glucose concentrations, and other endocrine factors (Pro-insulin, C-Peptide, Estrogen, triglycerides) in the pathogenesis of Type 2 diabetes and cardiovascular disease. Findings from this pilot study will inform public health recommendations for food packaging and provide much needed experimental evidence as to whether BPA poses any public health risk.

ELIGIBILITY:
Inclusion Criteria:

* BMI = 18.5-35
* Age 18-50 years
* Non-smoking
* English speaking

Exclusion Criteria:

* History of infertility
* Type 2 or Type 1 diabetes
* Cardiovascular disease, or any other metabolic disease/complication
* Hypertension (systolic blood pressure ≥140, diastolic blood pressure ≥90) assessed by sphygmomanometer
* History of major psychiatric illness, drug abuse, or unsafe dieting practices
* History of bariatric surgery
* Pregnant women or women expecting or trying to become pregnant
* Participating in other studies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Glucose at 180 Minutes | 9 samples over 3 hours at time minutes 0 (baseline), 15, 30, 45, 60, 90, 120, 180
  Glucose concentrations will be assessed before and in response to a 75 gram Oral Glucose Tolerance Test

SECONDARY OUTCOMES:
Change From Baseline Insulin at 180 Minutes | 9 samples over 3 hours at time minutes 0 (baseline), 15, 30, 45, 60, 90, 120, 180
  Insulin concentrations will be assessed before and in response to a 75 gram Oral Glucose Tolerance Test
Change From Baseline Estrogen at 180 Minutes | 9 samples over 3 hours at time minutes 0 (baseline), 15, 30, 45, 60, 90, 120, 180
  Estrogen concentrations will be assessed before and in response to a 75 gram Oral Glucose Tolerance Test
Change From Baseline C-Peptde at 180 Minutes | 9 samples over 3 hours at time minutes 0 (baseline), 15, 30, 45, 60, 90, 120, 180
  C-Peptide concentrations will be assessed before and in response to a 75 gram Oral Glucose Tolerance Test
Change From Baseline Pro-Insulin at 180 Minutes | 9 samples over 3 hours at time minutes 0 (baseline), 15, 30, 45, 60, 90, 120, 180
  Pro-Insulin concentrations will be assessed before and in response to a 75 gram Oral Glucose Tolerance Test
Change From Baseline Triglycerides at 180 Minutes | 9 samples over 3 hours at time minutes 0 (baseline), 15, 30, 45, 60, 90, 120, 180
  Triglyceride concentrations will be assessed before and in response to a 75 gram Oral Glucose Tolerance Test

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hagobian, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data in this pilot study